CLINICAL TRIAL: NCT01196858
Title: Duration of Untreated Psychosis (DUP) and Pathways to Care in Patients With First- and Multiple Episodes of Psychosis in Nordland - a Study of the Components of DUP in a Rural Mental Health System
Brief Title: Duration of Untreated Psychosis (DUP) and Pathways to Care in Nordland
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/1426(REK)
Record Dates: First submitted 2010-09-06; First posted 2010-09-09 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Schizophrenia and Disorders With Psychotic Features; Affective Psychosis, Bipolar; Psychoses
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Bipolar Disorder; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
During the 1990s, evidence began to emerge of the long duration of untreated illness prior to receiving treatment for patients with psychotic disorders. Studies across the world on first episode psychosis have consistently found an average of 1 - 2 years between the onset of psychotic symptoms and the start of treatment. Lengthy treatment delay has immediate implications such as unnecessary distress for patients and families, and may also compromise potential recovery when treatment is initiated.By understanding how and why substantial delays occur the investigators may be able to better design interventions to facilitate better earlier treatment. The components of DUP can be conceptualised as comprising 3 distinct intervals: help-seeking delay, referral delay and delay in mental health services. In this study the primary aim is to establish the level of DUP in nordland, and explore the components of this variable. Help-seeking delay will be investigated by interviewing patients presenting at the central mental health hospital in Nordland about their psychosis onset and pathways to care. Referral delay will be investigated by a questionnaire about the referral pratices among GPs in Nordland. Delays in mental health services will be investigated by focus group interviews with leaders and professionals at the 7 community mental health centers in Nordland. This knowledge is believed to be crucial for developing services that can reduce DUP and give this patient population earlier access to adequate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any patient presenting with a possible psychotic illness (including schizophrenia, affective psychosis and drug-related psychosis, but excluding organic psychosis).
* Understands and speaks norwegian

Exclusion Criteria:

* Severe learning disability

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study is a naturalistic cohort study. All patients registrered in a 3 year period with the acute and/or rehabilitation units will be invited to participate.
  The eight units (acute and rehabilitation) will be able to provide a potential sample size of 150 participants over the 3-year period of the study. We are confident of minimal attrition and assume that we will achieve at least 85% follow up. This means that we can expect to have collected data on approximately 120 people.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Duration of untreated psychosis | retrospective, lifetime
  Nottingham Onset Schedule

CONTACTS AND LOCATIONS:
Overall Officials: Knut W. Soergaard, PhD, Principal Investigator — Nordlandssykehuset HF
Locations (1):
- Nordland Hospital Trust, Bodø, Bodoe, Norway